CLINICAL TRIAL: NCT04400955
Title: A Prospective Cross-sectional Study Analysing the Utility of Novel Tablet-based Audiometry and an Interactive Web-based Hearing App as Screening Tools for Drug-induced Ototoxicity in Adult Cystic Fibrosis
Brief Title: A Study of Web and Tablet-based Interactive Audiometry in Adults With CF
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18/SC/0057
Record Dates: First submitted 2020-02-13; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Hearing Loss, Sensorineural; Cystic Fibrosis
MeSH Terms: conditions — Hearing Loss, Sensorineural; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood for genomic DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Audiometry tablet diagnostic tool and web-based test — as above

SUMMARY:
Adults with CF regularly receive anti-infective therapy that can result in impaired hearing. Recent studies have identified that up to 50% of adults with CF have hearing loss with resulting significant impact on quality of life. At present, however, there is no national recommendation to screen for hearing loss within adult CF.

Formal hearing tests are costly, require specialist staff and equipment and require further outpatient visits resulting in significant impact on health, social and financial resource.

We propose to analyse over a 12 month period at two adult cystic fibrosis centres in London whether outpatient tablet based audiometry testing and web-based hearing apps are able to accurately screen for ototoxicity in adults with CF, and whether these methods of screening are acceptable. The results of this study will aim to streamline audiometry screening to improve detection rates, reduce cost of healthcare, enable equity in service delivery, and minimize disruption to the patient's social and work-life using smart technology.

DETAILED DESCRIPTION:
Through a prospective multi-centre cross-sectional study, the utility of outpatient tablet-based audiometry (Shoebox MD, Clearwater Medical Ltd) and a novel interactive web-based hearing app developed in collaboration with the Dyson School of Audio design engineering, Imperial College (Project: 3D Tune-in) will be compared to standard sound-booth extended high-frequency audiometry performed by an audiologist and a validated ototoxicity screening questionnaire (HHIA). 200 adults with CF presenting either to the Specialist Adult Cystic Fibrosis Centre at the Royal Brompton and Harefield Foundation Trust or Kings College Hospital NHS Foundation Trust will be prospectively recruited to the study over a 12-month period. Blood samples for genomic DNA isolation will additionally be taken for all participants for mitochondrial DNA sequencing.

Hypothesis:

Tablet-based audiometry is a valid reliable tool to screen for drug-induced hearing loss in adults with CF.

Blinding:

- Audiologists performing standard sound-booth extended high-frequency audiometry will be blinded to results of tablet-based audiometry and web-based hearing app results.

Outcome measures:

* Warble-tone thresholds will be analysed through both tablet and standard extended high-frequency audiometry.
* Interclass correlation coefficient (ICC) with a 95% confidence interval will be used as a measure of reliability.
* Sensitivity, specificity and negative predictive value will be analysed to determine utility of tablet based audiometry, web-based hearing app, standardised hearing questionnaires and mitochondrial mutation screening to identify ototoxicity in adults with CF.
* Logistic regression modelling (complex statistical modelling) will be used to determine risk factors for developing hearing loss within adult CF.
* 7-point Likert scale questionnaires will be used to evaluate patient satisfaction, perceived usefulness and usability of tablet audiometry, web-based app hearing testing and formal audiometry.

ELIGIBILITY:
Inclusion Criteria:

* All patients >16 years old under adult cystic fibrosis unit at Royal Brompton or King's college cystic fibrosis centres.

Ability to provide informed consent to participate in the study (written and witnessed).

Exclusion Criteria:

* • Inability of patient to provide informed consent.

  * Patients with previously diagnosed visual impairment (due to web-based and tablet-based hearing app)
  * Established hearing loss with hearing aids in use (due to increased complexity of hearing tests required)
  * Inability to attend audiology outpatient appointments due to state of health.
  * Pregnancy (due to potential for reversible hearing loss during pregnancy affecting study reliability)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with Cystic Fibrosis at Royal Brompton and Kings hospital London.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Intraclass correlation coefficient with 95% CI | Through study completion, an average of 1 year
  Reliability of tablet audiometry compared to gold-standard

SECONDARY OUTCOMES:
Sensitivity, specificity of audiology screening tools | Through study completion, an average of 1 year
  as above
Logistic regression modeling to identify risk factors for sensorineural hearing loss in adults with CF | Through study completion, an average of 1 year
  as above

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Anand Shah, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and data available on request.
Supporting Information: Study Protocol, CSR
Time Frame: Available on completion of study on request
Access Criteria: Available on completion of study on request